CLINICAL TRIAL: NCT03363295
Title: Evaluation and Comparison of Macular and Choroidal Thickness After Intracameral Moxifloxacin for Prevention of Postcataract Endophthalmitis
Brief Title: Evaluation of Macular Changes After Intracameral Moxifloxacin for Prevention of Endophthalmitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pessoa Cavalcanti Lira, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2017-11-25; First posted 2017-12-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Endophthalmitis; Macula Edema; Cataract
Keywords: endophthalmitis
MeSH Terms: conditions — Endophthalmitis; Cataract | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the patients and the investigator will be masked. The cataract surgeon won't be.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intracameral moxifloxacin (Experimental): Injection of 0,03ml of moxifloxacin in the anterior chamber following phacoemulsification surgery
  Interventions: Drug: Moxifloxacin Injection
- No - Intracameral moxifloxacin (No Intervention): This group won't receive any prophylaxis after phacoemulsification surgery

INTERVENTIONS:
Drug: Moxifloxacin Injection — One group will receive moxifloxacin injection (0,03ml) in the anterior chamber by the end of phacoemulsification surgery
  Arms: Intracameral moxifloxacin

SUMMARY:
The objective of this study is to evaluate the macular and choroidal thickness of patients submitted to intracameral moxifloxacin during the phacoemulsification surgery for endophthalmitis prophylaxis.

The investigators propose a randomized clinical trial double-blind. The patients will be divided into two groups: one will receive intracameral moxifloxacin injection during phacoemulsification surgery and the other won't.

Both Spectral Domain - Optical Coherence Tomography (SD-OCT) and Enhanced Depth Imaging - Optical Coherence Tomography (EDI-OCT) will be performed for each patient pre-operatively and on the 30th and 60th postoperative days.

After collecting, the data will be compared to evaluate if there was any difference in the macular thickness and choroidal thickness between the two groups.

DETAILED DESCRIPTION:
Title:

Evaluation and Comparison of Macular and Choroidal Thickness after Intracameral Moxifloxacin for Prevention of Postcataract Endophthalmitis

Purpose:

The objective of this study is to evaluate if the using of intracameral moxifloxacin cause changes in macular and choroidal thickness.

Methods:

A randomized clinical trial will be conducted in the Hospital of Clinics at State University of Campinas (UNICAMP). The patients that will be submitted to phacoemulsification surgery will be divided into two groups. The first group will receive 0,03ml intracameral moxifloxacin after phacoemulsification surgery, while the second group won't receive any antibiotics intracamerally. Both groups will apply eyedrops as usual in the postoperative.

The investigators will evaluate those patients blindly. Each patient will be examined using Spectral Domain - Optical Coherence Tomography (SD-OCT) and Enhanced Depth Imaging - Optical Coherence Tomography (EDI-OCT), in the pre-operative, at the 30th postoperative and at the 60th postoperative. The data will be collected regarding macular central thickness and choroidal thickness.

The exclusion criteria will be:

* Patients who had any macular changes prior to the surgery (including epiretinal membrane, macular edema, drusen or any other)
* diabetic patients
* patients who had any complications during the cataract surgery
* patients who refuse to participate in the trial, or refuse to sign the consent form

After collecting data, the two groups will be compared regarding changes in macular thickness and choroidal thickness from the pre-operative, the 30th and the 60th postoperative.

The investigators expect that there will be no statistical difference between groups

ELIGIBILITY:
Inclusion Criteria:

* Any patients that will be submitted to phacoemulsification surgery in the Hospital de Clinicas of State University of Campinas (BRAZIL)
* Patients over 18 years old
* Patients who are able to perform SD-OCT
* Patients who sign the consent form

Exclusion Criteria:

* Diabetic patients
* Patients with any macular changes prior to the surgery (epiretinal membranes, age macular disease, macular edema...)
* Patients who had any complication during phacoemulsification surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Macular Thickness | Change from baseline, 30th day postoperative and 60th day postoperative
  Comparison of change in macular thickness using Spectral Domain - Optical Coherence Tomography

SECONDARY OUTCOMES:
Change of Choroidal Thickness | Change from baseline, 30th day postoperative and 60th day postoperative
  Comparison of change in macular thickness using Enhanced Depth Imaging - Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mathias V Mélega, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Hospital das Clínicas da UNICAMP, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira BG, Cardoso da Silva I, Melega MV, Nascimento MA, Cavalcanti Lira RP, Leite Arieta CE, Alves M. Macular and choroidal thickness after intracameral moxifloxacin for prevention of postcataract endophthalmitis. J Cataract Refract Surg. 2021 Jan 1;47(1):40-45. doi: 10.1097/j.jcrs.0000000000000365. PMID 32818353